CLINICAL TRIAL: NCT02126306
Title: Beta Glucosylceramide for Treatment of Non Alcoholic Steatohepatitis
Brief Title: Beta Glucosylceramide for Treatment of NASH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YI1958
Record Dates: First submitted 2014-04-09; First posted 2014-04-30 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2006-01

CONDITIONS: Compliance Behavior
MeSH Terms: conditions — Patient Compliance | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline administered orally daily as a placebo
  Interventions: Drug: Placebo
- Beta Glucosylceramide (Active Comparator): Beta glucosylceramide administered orally daily
  Interventions: Drug: Beta Glucosylceramide

INTERVENTIONS:
Drug: Beta Glucosylceramide — Beta Glucosylceramide
  Arms: Beta Glucosylceramide
Drug: Placebo — normal saline
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
Oral administration of betaglucosylceramide was shown effective in reducing inflammation in animal models and was found safe in humans.

DETAILED DESCRIPTION:
Patients with NASH to receive the treatment versus placebo for 40 weeks followed by a liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven NASH

Exclusion Criteria:

* Other therapies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, M.D., Study Director — Hadassah Medical Organization

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
  Beta Glucosylceramide: Beta Glucosylceramide
  placebo: placebo
- Beta Glucosylceramide: Beta Glucosylceramide 7.5 mg
  Beta Glucosylceramide: Beta Glucosylceramide
  placebo: placebo
Period: Overall Study
Arm/Group | Placebo | Beta Glucosylceramide
Started | 10 | 13
Completed | 10 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Beta Glucosylceramide: Beta Glucosylceramide
  Beta Glucosylceramide: Beta Glucosylceramide
  placebo: placebo
- Total: Total of all reporting groups
Arm/Group | Placebo | Beta Glucosylceramide | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  Israel | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease of 2 Points in the Non-Alcoholic Fatty Liver Disease Activity Score (NAS) Analysis is Per Protocol
Description: Number of Participants who had a decrease of 2 points in the Non-Alcoholic Fatty Liver Disease Activity Score (NAS) from baseline at 40 weeks per protocol analysis. The score is performed on the liver biopsy before and after treatment. The total score is used with a range from 4-16. A decrease in the total score by 2 points or more is considered an improvement, while an increase in the total score by 2 points or more is considered deterioration. No use of subscales for the data analysis was made.
  Allparticipants in both arms who showed a decrease of 2 points or more in the Non-Alcoholic Fatty Liver Disease Activity Score are conisdered as responders. Only values quantifying data that were actually measured and analyzed are included.
Time Frame: Total score from baseline compared with week 40.
Measure: Number; unit: participants
Groups:
- Placebo: Placebo
  Beta Glucosylceramide: Beta Glucosylceramide
  placebo: placebo NAS score
- Beta Glucosylceramide: Beta Glucosylceramide
  Beta Glucosylceramide: Beta Glucosylceramide
  placebo: placebo NAS score
Arm/Group | Placebo | Beta Glucosylceramide
Number analyzed (Participants) | 10 | 13
participants | 10 | 13

ADVERSE EVENTS:
Time Frame: 40 weeks
Arm/Group | Placebo | Beta Glucosylceramide
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 0/10 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No